CLINICAL TRIAL: NCT05941728
Title: Persea Americana for Total Health (PATH)-2
Acronym: PATH-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Hannah Holscher, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22788
Record Dates: First submitted 2023-06-27; First posted 2023-07-12 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Overweight and Obesity
Keywords: Avocado; Gastrointestinal microbiome; Bile acid profile; Inflammation; Thinking; Glycemia
MeSH Terms: conditions — Overweight; Obesity; Inflammation | interventions — Oils; Dietary Fiber

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Avocado (Experimental): The experimental treatment will contain an avocado. Avocados will be consumed daily for 4 weeks.
  Interventions: Other: Avocado
- Fiber + Oil (Active Comparator): The active comparator will have a snack that mimics the fiber and fatty acid composition found in avocados and will be consumed daily for 4 weeks.
  Interventions: Other: Oil + Fiber
- Standard American Diet (Sham Comparator): The sham comparator contains foods and beverages of a standard American diet and will be consumed daily for 4 weeks.
  Interventions: Other: Average American Diet

INTERVENTIONS:
Other: Avocado — The intervention treatment will contain avocado
  Arms: Avocado
Other: Oil + Fiber — The active comparator will contain a snack with oils and fibers that mimic an avocado
  Arms: Fiber + Oil
Other: Average American Diet — The sham comparator will contain foods/beverages that mimic a standard American Diet
  Arms: Standard American Diet

SUMMARY:
The goal of this clinical trial is to learn about the effects of avocado consumption on gastrointestinal health in adults with overweight and obesity. The main questions is aims to answer are:

How does avocado consumption affect the gut microbiome? How does avocado consumption affect thinking? Are there connections between the microbiome and cognition? Participants will be asked to eat provided meals with and without avocados for three 4-week periods. At the end of each 4-week period, participants will be asked to provide stool samples and complete computer games that assess thinking and memory.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 25 and 74 years old
* BMI ≥ 25 kg/m2
* Ability to drop off fecal sample within 15 minutes of defecation
* 20/20 or corrected vision

Exclusion Criteria:

* Avocado allergy or intolerance
* Food allergies or intolerances
* Prior diagnosis of liver or gastrointestinal disease (primary biliary cirrhosis or gallbladder disease, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers), diabetes, hepatitis, HIV, or cancer
* Women that are pregnant, have given birth in the previous 12 months or are lactating
* Individuals that smoke, use tobacco, abuse drugs, or consume > 2 alcoholic beverages per day.
* > 5% weight change in the past month or > 10% change in the past six months
* Oral antibiotics during the previous 6 weeks.
* Currently taking lipid-lowering medications, oral hypoglycemic agents, or insulin.
* History of malabsorptive or restrictive bariatric surgeries (e.g., gastric bypass, sleeve gastrectomy, adjustable gastric band) or gall bladder removal surgery.
* Are unable to consume the experimental meals/snacks.
* Allergic to latex
* Concurrent enrollment in another dietary, exercise, or medication study

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Fecal microbial species | 4 weeks
  Feacalibacterium spp., bacteria capable of producing SCFA and secondary bile acid synthesis measured using metagenomic sequencing
Fecal microbial genes | 4 weeks
  Microbial genes involved in short-chain fatty acids and secondary bile acid synthesis measured using metagenomic sequencing
Concentration of fecal bile acids | 4 weeks
  Fecal bile acid concentrations using HPLC in avocado and active comparator vs. control,
Concentration of fecal SCFA | 4 weeks
  Fecal SCFA concentrations using GC-MS in avocado and active comparator vs. control,

SECONDARY OUTCOMES:
Cognitive function | 4 weeks
  Neuropshycological function as measured by a clinical cognitive task battery.
Subjective gastrointestinal tolerance via questionnaire | 4 week
  Ratings of gastrointestinal symptoms (ease of stool passage, frequency of stools, abdominal pain, bloating, burping, flatulence, nausea, reflux, rumblings assessed using questionnaires
Digestive health using stool records/Bristol Stool Scale | 4 week
  Ratings of stool consistency using Bristol Stool Scale

OTHER OUTCOMES:
Fecal microbiome | 4 weeks
  Relative abundance of microbial genes, genera, and community structure measured using metagenomic sequencing of extracted fecal DNA to compare abundances between avocado, active comparator, and control.
Inflammation | 4 weeks
  LPS-binding protein, a marker of inflammation will be measured using ELISA. (Blood samples)
Intestinal permeability | up to 4 weeks
  Intestinal permeability will be measured using a orally ingested sugar substitutes. 24-hour urinary appearance of the sugars will be quantified using GC-MS.
Fecal metabolites | 4 weeks
  Proteolytic metabolites will be measures in fecal samples using GC-MS
Fecal pH | 4 weeks
  Fecal pH will be measured using a pH meter

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Holscher, PhD, RD, Principal Investigator — University of Illinois Urbana Champaign
Locations (1):
- University of Illinois, Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No